CLINICAL TRIAL: NCT01920906
Title: Comparative Analysis of Small and Large Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Jaehwan Kim, Clinical Scholar, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JWK-0816
Record Dates: First submitted 2013-08-06; First posted 2013-08-12 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; Korean; Healthy Volunteers
MeSH Terms: conditions — Psoriasis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biopsy and blood tests (Experimental): All subjects will undergo a skin biopsy and blood tests
  Interventions: Procedure: Skin biopsy and blood test

INTERVENTIONS:
Procedure: Skin biopsy and blood test — Analysis of histology and gene expression in affected and unaffected skin

SUMMARY:
Psoriasis is a chronic, debilitating skin disorder with an estimated prevalence of 2%. Psoriatic skin lesions start with initial pinhead-sized macules and then coalesce into plaques of varying sizes. Despite the great strides in the studies for psoriasis, it is still unclear why psoriatic skin lesions start with small macules and then spread peripherally.

To study peripheral spreading of psoriasis, investigators plan to study small plaque psoriasis in comparison to large plaque psoriasis in the Korean population. Large plaque psoriasis is the most common form of psoriasis, seen in approximately 90% of all psoriasis participants. Large psoriatic plaques are >5 cm in size and localize to the extensor aspects of the elbows, knees, scalp, and genital area. On the other hand, small plaque psoriasis is the common or typical form of psoriasis that occurs particularly in Korea and other Asian countries. Korean small plaque psoriasis, even when chronic, remains <2 cm in size and is widely distributed on the upper trunk and proximal extremities.

Investigators hypothesize that the expression of immune-related genes are different between small and large plaque psoriasis. The study of a genetically homogeneous cohort, characterized by the relatively high prevalence of small plaque psoriasis in the Korean population, may filter out spurious signals while allowing for significant associations to emerge from a relatively low number of participants.

By comparing small and large plaque psoriasis, it is expected this study could lead to new understandings of the mechanisms involved in spreading of psoriatic plaques and provide new insights into psoriasis development.

DETAILED DESCRIPTION:
Psoriasis is a common chronic skin disorder with an estimated prevalence in populations of approximately 2%. Psoriatic skin lesions start with initial pinhead-sized macules and then coalesce into plaques of varying sizes in diameter from one to several centimeters.

Despite the great strides in the studies for psoriasis, it is still unclear why psoriatic skin lesions start with small macules and then spread peripherally. The occurrence of psoriasis is thought to be the pathological consequence of an exaggerated immune response as activated T cells, monocytes, neutrophils, and dendritic cells produce inflammatory cytokines that drive the additional recruitment of inflammatory cells, further elaboration of proinflammatory mediators, and the proliferation of keratinocytes. However, pathogenetic mechanism for peripheral spreading of psoriasis needs to be further elucidated.

To study peripheral spreading of psoriasis, investigators plan to study "small plaque psoriasis" and compare it to "large plaque psoriasis" in the Korean population.

Psoriasis vulgaris, so-called "large plaque psoriasis", is the most common form of psoriasis, seen in approximately 90% of all psoriasis patients. Red, scaly, symmetrically distributed plaques are usually larger than 5 cm in diameter and characteristically localized to the extensor aspects of the extremities, particularly the elbows and knees, along with scalp, lower lumbosacral, buttocks, and genital involvement. Approximately 1/4 to 1/3 of large plaque psoriasis participants have involvement of over 5% of their body surface area (BSA), and disease of this extent is frequently painful and physically and/or socially debilitating to a degree comparable with other chronic medical conditions.

On the other hand, "small plaque psoriasis" is the common or typical form of psoriasis that occurs in adults particularly in Korea and other Asian countries. Korean small plaque psoriasis, even when chronic, remain <2 cm in size and widely distributed on upper trunk and proximal extremities. Small plaque psoriasis is less severe than large plaque psoriasis, as it usually responds to phototherapy and more potent therapies are rarely needed.

It is also noteworthy that there are well-known human leukocyte antigen (HLA) differences in Caucasians in comparison with Asian participants with psoriasis, and a unique HLA haplotype has been described in Korean participants with psoriasis. Furthermore, an allele of an HLA-related gene, known as major histocompatibility complex I chain-related gene A, is known as a susceptibility marker in Korean and Chinese participants with psoriasis, but not in Spanish participants.

For a more comprehensive analysis of the difference between small and large plaque psoriasis, investigators plan to compare these two different types of psoriasis only in the Korean population. The study of a genetically homogeneous cohort, characterized by the relatively high prevalence of small plaque psoriasis in the Korean population, may filter out spurious signals while allowing for significant associations to emerge from a relatively low number of participants. By comparing Korean psoriasis participants in two geographically separated locations (Seoul, Korea vs. New York, NY, USA), it will also be interesting to understand the interactions between genetics and the environment that are still not well defined.

It is anticipated this study could lead to new understanding of the mechanisms involved in the spreading of psoriatic plaques and provide new insight into psoriasis pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Korean (defined as being Korean and both parents are Korean)
* History of small and/or large plaque psoriasis, for at least six months
* At least 18 years of age
* No treatment with topical steroids or vitamin D analogues for at least 2 weeks prior to entering the study.
* No treatment with systemic therapies, including phototherapy, acitretin, cyclosporine, methotrexate and biologics 4 weeks prior to entering the study. Among biologics, Ustekinumab (Stelara®) requires a longer washout period of 12 weeks.

Exclusion Criteria:

* Erythrodermic, or pustular psoriasis as the sole or predominant form of psoriasis.
* Photosensitizing illnesses such as lupus, polymorphous light eruption, or any disease known to be worsened by UV light exposure.
* History of malignant melanoma.
* Pregnancy.
* Immunocompromising diseases such as HIV infection.
* Inflammatory diseases such as but not limited to Crohn's Disease, Multiple Sclerosis, Rheumatoid Arthritis, Hashimoto's Disease.
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data. Participants taking medications that induce photosensitivity may be included after careful review.
* Poorly controlled medical conditions of any kind.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the RT-PCR measurement of IL-17 in lesional psoriasis skin samples collected from patients in Korea. | 2 years
  The primary outcome measure is the expression of IL-17 (the pivotal immune related molecule in psoriasis pathogenesis) in lesional psoriatic skin samples collected from patients in Korea. The expression of IL-17 is measured by Reverse transcription polymerase chain reaction (RT-PCR) and normalized to the expression of housekeeping gene (human acidic ribosomal protein [hARP]). The unit of outcome measure is log2(IL-17 expression/hARP expression).

SECONDARY OUTCOMES:
The secondary outcome measure is the RT-PCR measurement of IL-17 in lesional psoriasis skin samples collected from patients at The Rockefeller Hospital, New York. | 2 years
  The secondary outcome measure is the expression of IL-17 (the pivotal immune related molecule in psoriasis pathogenesis) in lesional psoriatic skin samples collected from patients at The Rockefeller Hospital, New York. The expression of IL-17 is measured by Reverse transcription polymerase chain reaction (RT-PCR) and normalized to the expression of housekeeping gene (human acidic ribosomal protein [hARP]). The unit of outcome measure is log2(IL-17 expression/hARP expression).

CONTACTS AND LOCATIONS:
Overall Officials: Jaehwan Kim, MD PhD, Principal Investigator — Rockefeller Univesrity
Locations (1):
- The Rockefeller University, New York, New York, United States